CLINICAL TRIAL: NCT00697112
Title: Surveillance Registry Of Sirolimus Use In Recipients Of Kidney Allograft From Expanded Criteria Donors (ECD)
Brief Title: Study Evaluating The Use Of Sirolimus In Recipients Of Kidney Allografts From Expanded Criteria Donors (ECD)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0468H-102385; B1741025
Record Dates: First submitted 2008-06-10; First posted 2008-06-13 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-12

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Non interventional. Sirolimus administered by Principal Investigator per standard practice and labeling.
  Other Names: Rapamune

SUMMARY:
The purpose of this observational study is to examine the clinical outcomes of the use of sirolimus as base therapy in kidney allograft recipients from Expanded Criteria Donors (ECD) under conditions of routine clinical practice. The primary objective is to identify the current criteria/reasons to use sirolimus as base therapy in this selected population and define and understand the emerging patterns of immunosuppressive treatment with sirolimus.

DETAILED DESCRIPTION:
pilot study

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients who received a renal transplant (primary, secondary, tertiary, etc.) without pancreas, from Expanded Criteria Donors (ECD), 3 months prior and no later than 1 year at the time of study enrollment.
* Patients who provided informed consent.
* Patients without sirolimus as base therapy.

Exclusion Criteria:

* Patients who are unwilling or unable to provide informed consent or who lack a legal guardian or designee able to provide consent on their behalf.
* Patients who are unable to complete the study.
* Patients who are participating in another clinical trial during the last 6 months.
* Pregnant or lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney allograft recipients
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Argentina (5):
  - Pfizer Investigational Site, Caba, Buenos Aires
  - Pfizer Investigational Site, Barrio General Paz, Córdoba Province
  - Pfizer Investigational Site, Santa Fe, Santa Fe Province
  - Pfizer Investigational Site, San Miguel de Tucumán, Tucumán Province
  - Pfizer Investigational Site, Córdoba

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0468H-102385&StudyName=Study%20Evaluating%20The%20Use%20Of%20Sirolimus%20In%20Recipients%20Of%20Kidney%20Allografts%20From%20Expanded%20Criteria%20Donors%20%28ECD%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus: Participants who had kidney transplant from expanded criteria donors (ECD) and received sirolimus (Rapamune) as base therapy in immunosuppressive regimen according to the standard clinical practice as determined by the physician, were followed up for 1 year. The term ECD refers to kidneys from deceased donors who were either 60 years and older or aged 50 to 59 years with 2 of 3 conditions (serum creatinine level greater than [>] 1.5 milligram per deciliter [mg/dL], cerebrovascular accident as cause of death or history of hypertension).
Period: Overall Study
Arm/Group | Sirolimus
Started | 53
Met the Inclusion Criteria | 52
Completed | 43
Not Completed | 10
Not completed — Adverse Event | 8
Not completed — Lost to Follow-up | 1
Not completed — Did not meet inclusion criteria | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had received at least 1 dose of Rapamune and were subsequently interrogated.
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Main Reason for the Use of Sirolimus (Rapamune) Therapy
Description: The study employ a questionnaire which included different clinical criteria to determine the main medical reason for the introduction of sirolimus (Rapamune) therapy after renal transplant. The physician responsible selected the one that was considered the main reason for introduction of sirolimus (Rapamune) as base immunosuppressive therapy.
Time Frame: Baseline
Population: Intention-to-Treat (ITT) population included all participants who were treated with Rapamune for at least 4 or 5 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
percentage of participants
  Calcineurin inhibitor (CNI) nephrotoxicity | 40.38 [27.01 to 54.90]
  Chronic allograft nephropathy | 25.00 [14.03 to 38.95]
  Metabolic disorders | 5.77 [1.21 to 15.95]
  To prevent chronic allograft nephropathy | 5.77 [1.21 to 15.95]
  Tumoral history | 5.77 [1.21 to 15.95]
  Virological status | 5.77 [1.21 to 15.95]
  Delay graft function | 3.85 [0.47 to 13.21]
  Expanded criteria donor characteristics | 3.85 [0.47 to 13.21]
  Diarrhea | 1.92 [0.05 to 10.26]
  To prevent CNI nephrotoxicity | 1.92 [0.05 to 10.26]

2. Secondary Outcome: Probability of Graft Survival
Description: Graft survival was considered in participants who did not experience graft failure. Graft failure was determined by return to dialysis for a period of at least 12 weeks with no return of function, or graft loss whichever occurred sooner.
Time Frame: Month 12
Population: ITT population included all participants who were treated with Rapamune for at least 4 or 5 weeks.
Measure: Number (95% Confidence Interval); unit: probability of graft survival
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
probability of graft survival | 1 [NA to NA] — Confidence interval was not calculated as none of the participants had graft failure.

3. Secondary Outcome: Probability of no Acute Rejection
Description: Diagnosis of acute rejection was made via kidney biopsy. Categorization of biopsies with suspected acute rejection was based on histological findings using updated 1997 Banff criteria: Grade 1A: significant interstitial infiltration (greater than [>] 25 percent [%] of parenchyma affected) and foci of moderate tubulitis (5-10 cells/tubular cross section), Grade 1B: significant interstitial infiltration (>25% of parenchyma affected) and severe tubulitis (>10 mononuclear cells/tubular cross section), Grade 2A: mild-moderate intimal arteritis, Grade 2B: severe intimal arteritis comprising >25% of the luminal area and Grade 3: transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells. Probability of no acute rejection throughout the sirolimus (Rapamune) therapy was estimated using Kaplan-Meier method.
Time Frame: Month 12
Population: ITT population included all participants who were treated with Rapamune for at least 4 or 5 weeks.
Measure: Number (95% Confidence Interval); unit: probability of no acute rejection
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
probability of no acute rejection | 0.960 [0.908 to 1]

4. Secondary Outcome: Probability of Participant Survival
Description: Participant's survival defined as participant living with or without a functioning graft. Probability of participant survival throughout the sirolimus (Rapamune) therapy was estimated using Kaplan-Meier method.
Time Frame: Month 12
Population: ITT population included all participants who were treated with Rapamune for at least 4 or 5 weeks.
Measure: Number (95% Confidence Interval); unit: probability of participant survival
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
probability of participant survival | 0.979 [0.938 to 1]

5. Secondary Outcome: Average Dose of Immunosuppressive Drugs Administered
Description: Immunosuppressive drugs administered included cyclosporin A (CsA) administration based on monitoring of plasma trough levels (C0), CsA administration based on monitoring of plasma levels 2-hours after CsA dose (C2), tacrolimus, and sirolimus (Rapamune).
Time Frame: Baseline, Week 1 or 2, 4 or 5, 12 or 13, 24 or 25, 52 or 53
Population: ITT population. N(number of participants analyzed)=participants evaluable for this measure. n=participants evaluable at given time point for specified immunosuppressive. Results not reported for CsA C0 at Week 1/2, 12/13, 24/25; CsA C2 at Week 1/2, 4/5, 12/13, 24/25, 52/53; sirolimus at baseline as no participants evaluable at those time points.
Measure: Mean (Standard Deviation); unit: milligram per day
Arm/Group | Sirolimus
Number analyzed (Participants) | 47
milligram per day
  Baseline: CsA (C0) (n=3) | 200.00 (50.00)
  Baseline: CsA (C2) (n=3) | 306.67 (83.27)
  Baseline: Tacrolimus (n=40) | 5.74 (2.73)
  Week 1 or 2: Tacrolimus (n=12) | 4.79 (2.28)
  Week 1 or 2: Sirolimus (n=44) | 2.43 (0.84)
  Week 4 or 5: CsA (C0) (n=1) | 150.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Week 4 or 5: Tacrolimus (n=6) | 3.67 (2.93)
  Week 4 or 5: Sirolimus (n=42) | 2.52 (0.80)
  Week 12 or 13: Tacrolimus (n=4) | 4.00 (2.55)
  Week 12 or 13: Sirolimus (n=47) | 2.45 (0.94)
  Week 24 or 25: Tacrolimus (n=2) | 4.21 (3.95)
  Week 24 or 25: Sirolimus (n=46) | 2.35 (0.99)
  Week 52 or 53: CsA (C0) (n=1) | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Week 52 or 53: Tacrolimus (n=1) | 3.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Week 52 or 53: Sirolimus (n=36) | 2.05 (0.89)

6. Secondary Outcome: Average Blood Level of Immunosuppressive Drugs Administered
Description: as for outcome 5
Time Frame: Baseline, Week 1 or 2, 4 or 5, 12 or 13, 24 or 25, 52 or 53
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Sirolimus
Number analyzed (Participants) | 47
nanogram per milliliter (ng/mL)
  Baseline: CsA (C0) (n=3) | 144.00 (36.66)
  Baseline: CsA (C2) (n=3) | 580.67 (251.64)
  Baseline: Tacrolimus (n=40) | 7.82 (2.14)
  Week 1 or 2: Tacrolimus (n=12) | 8.12 (3.14)
  Week 1 or 2: Sirolimus (n=44) | 8.55 (3.83)
  Week 4 or 5: CsA (C0) (n=1) | 136.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Week 4 or 5: Tacrolimus (n=6) | 7.00 (5.60)
  Week 4 or 5: Sirolimus (n=42) | 7.81 (3.33)
  Week 12 or 13: Tacrolimus (n=4) | 5.42 (3.86)
  Week 12 or 13: Sirolimus (n=47) | 7.39 (2.25)
  Week 24 or 25: Tacrolimus (n=2) | 4.15 (1.91)
  Week 24 or 25: Sirolimus (n=46) | 7.75 (2.68)
  Week 52 or 53: CsA (C0) (n=1) | 86.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Week 52 or 53: Tacrolimus (n=1) | 2.40 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Week 52 or 53: Sirolimus (n=36) | 7.44 (2.54)

7. Secondary Outcome: Average Creatinine Clearance
Description: Creatinine clearance (CCr) is a measure of glomerular filtration rate (GMFR), an index of kidney function. CCr is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Normal values for healthy, young males are in the range of 100-135 milliliter per minute (mL/min) and for females, 90-125 mL/min. Creatinine clearance decreases with age. A low creatinine clearance rate indicates poor kidney function.
Time Frame: Baseline, Week 1 or 2, 4 or 5, 12 or 13, 24 or 25, 52 or 53
Population: ITT population included all participants who were treated with Rapamune for at least 4 or 5 weeks. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: milliliter per minute (mL/min)
Arm/Group | Sirolimus
Number analyzed (Participants) | 51
milliliter per minute (mL/min)
  Baseline (n=51) | 45.40 (19.00)
  Week 1 or 2 (n=49) | 50.56 (18.02)
  Week 4 or 5 (n=47) | 51.51 (21.45)
  Week 12 or 13 (n=48) | 50.95 (18.91)
  Week 24 or 25 (n=46) | 49.52 (19.77)
  Week 52 or 53 (n=38) | 53.24 (22.60)

8. Secondary Outcome: Average Proteinuria
Description: Proteinuria defined as the presence of an excess of serum proteins in the urine. Normal value of proteinuria is below 0.15 grams per 24 hours (g/24 hr).
Time Frame: Baseline, Week 1 or 2, 4 or 5, 12 or 13, 24 or 25, 52 or 53
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/24 hr
Arm/Group | Sirolimus
Number analyzed (Participants) | 29
g/24 hr
  Baseline (n=29) | 0.17 (0.20)
  Week 1 or 2 (n=24) | 0.19 (0.16)
  Week 4 or 5 (n=24) | 0.37 (0.60)
  Week 12 or 13 (n=25) | 0.48 (0.89)
  Week 24 or 25 (n=23) | 0.60 (1.16)
  Week 52 or 53 (n=18) | 0.45 (0.63)

9. Secondary Outcome: Percentage of Participants Who Prematurely Discontinued the Sirolimus (Rapamune) Therapy
Time Frame: Baseline up to Month 12
Population: ITT population included all participants who were treated with Rapamune for at least 4 or 5 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
percentage of participants | 15.38

10. Secondary Outcome: Percentage of Participants Who Prematurely Discontinued the Sirolimus (Rapamune) Therapy Due to Inefficacy
Time Frame: Baseline up to Month 12
Population: ITT population included all participants who were treated with Rapamune for at least 4 or 5 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
percentage of participants | 0

11. Secondary Outcome: Percentage of Participants Who Prematurely Discontinued the Sirolimus (Rapamune) Therapy Due to Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Participants who discontinued sirolimus (Rapamune) therapy prematurely due to AE were obliged to discontinue sirolimus (Rapamune) therapy permanently, are reported.
Time Frame: Baseline up to Month 12
Population: ITT population included all participants who were treated with Rapamune for at least 4 or 5 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
percentage of participants | 15.38

12. Secondary Outcome: Body Mass Index
Description: BMI was calculated as weight divided by height squared and measured as kilogram per square meter (kg/m^2).
Time Frame: Baseline, Week 1 or 2, 4 or 5, 12 or 13, 24 or 25, 52 or 53
Population: Safety population included all participants who had received at least 1 dose of Rapamune and were subsequently interrogated. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Sirolimus
Number analyzed (Participants) | 24
kg/m^2
  Baseline (n=24) | 24.48 (3.65)
  Week 1 or 2 (n=18) | 23.74 (3.69)
  Week 4 or 5 (n=24) | 24.94 (4.26)
  Week 12 or 13 (n=17) | 24.70 (3.99)
  Week 24 or 25 (n=17) | 25.01 (3.76)
  Week 52 or 53 (n=13) | 24.06 (3.16)

13. Secondary Outcome: Number of Participants With Body Temperature
Description: Body temperature was measured in degree Celsius. Each participants were classified into three different categories based on their body temperature: body temperature less than 35 degree Celsius = hypothermia, body temperature between 35 to 37.5 degree Celsius = feverless, and body temperature greater than 37.5 degree Celsius = fever.
Time Frame: Baseline, Week 1 or 2, 4 or 5, 12 or 13, 24 or 25, 52 or 53
Population: Safety population. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time points. Results for hypothermia not reported as none of the participants was found hypothermic.
Measure: Number; unit: participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 26
participants
  Baseline: Feverless (n=21) | 21
  Week 1 or 2: Feverless (n=26) | 26
  Week 4 or 5: Feverless (n=25) | 25
  Week 12 or 13: Feverless (n=17) | 16
  Week 12 or 13: Fever (n=17) | 1
  Week 24 or 25: Feverless (n=17) | 17
  Week 52 or 53: Feverless (n=14) | 14

14. Secondary Outcome: Blood Pressure
Description: Systolic and diastolic blood pressure (BP) was measured after the participant had rested in the supine position for at least 5 minutes with the participant's arm supported at the level of the heart, and recorded to the nearest millimeters of mercury (mmHg).
Time Frame: Baseline, Week 1 or 2, 4 or 5, 12 or 13, 24 or 25, 52 or 53
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sirolimus
Number analyzed (Participants) | 48
mmHg
  Baseline: Systolic BP (n=48) | 127.8 (15.8)
  Baseline: Diastolic BP (n=48) | 77.2 (11.7)
  Week 1 or 2: Systolic BP (n=48) | 125.7 (13.4)
  Week 1 or 2: Diastolic BP (n=48) | 77.6 (9.3)
  Week 4 or 5: Systolic BP (n=45) | 127.4 (19.8)
  Week 4 or 5: Diastolic BP (n=45) | 75.6 (9.6)
  Week 12 or 13: Systolic BP (n=47) | 131.4 (17.1)
  Week 12 or 13: Diastolic BP (n=47) | 79.3 (9.8)
  Week 24 or 25: Systolic BP (n=40) | 128.9 (18.9)
  Week 24 or 25: Diastolic BP (n=40) | 77.0 (9.9)
  Week 52 or 53: Systolic BP (n=37) | 127.5 (15.7)
  Week 52 or 53: Diastolic BP (n=37) | 77.8 (9.8)

15. Secondary Outcome: Pulse Rate
Time Frame: Baseline, Week 1 or 2, 4 or 5, 12 or 13, 24 or 25, 52 or 53
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Sirolimus
Number analyzed (Participants) | 31
beats per minute
  Baseline (n=26) | 74.0 (7.9)
  Week 1 or 2 (n=27) | 77.4 (7.2)
  Week 4 or 5 (n=31) | 77.2 (9.0)
  Week 12 or 13 (n=22) | 73.2 (9.7)
  Week 24 or 25 (n=22) | 75.3 (10.1)
  Week 52 or 53 (n=22) | 76.2 (9.2)

16. Secondary Outcome: Body Weight
Time Frame: Baseline, Week 1 or 2, 4 or 5, 12 or 13, 24 or 25, 52 or 53
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Sirolimus
Number analyzed (Participants) | 46
kilogram
  Baseline (n=46) | 70.78 (14.50)
  Week 1 or 2 (n=46) | 71.17 (13.76)
  Week 4 or 5 (n=45) | 70.87 (14.25)
  Week 12 or 13 (n=43) | 72.85 (13.11)
  Week 24 or 25 (n=37) | 72.18 (13.48)
  Week 52 or 53 (n=34) | 70.96 (13.77)

17. Secondary Outcome: Percentage of Participants With Physical Abnormalities
Description: Physical abnormalities included all the abnormalities related to general disorders and administration site conditions, gastrointestinal disorders, skin and subcutaneous tissue disorders, vascular disorders, investigations, infections and infestations, eye disorders, respiratory, thoracic and mediastinal disorders, nervous system disorders, musculoskeletal and connective tissue disorders, injury, poisoning and procedural complications, surgical and medical procedures, psychiatric disorders, neoplasms benign, malignant and unspecified (incl cysts and polyps), ear and labyrinth disorders, and congenital, familial and genetic disorders.
Time Frame: Baseline up to Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
percentage of participants | 69.23

18. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug.
Time Frame: Baseline up to Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
percentage of participants | 88.46

19. Secondary Outcome: Percentage of Participants With Serious Adverse Events
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
percentage of participants | 40.38

20. Secondary Outcome: Percentage of Participants With Clinically-Significant Electrocardiogram Abnormalities
Description: Standard 12-lead ECG was performed. ECG intervals included PR interval (time between the onset of atrial depolarization and the onset of ventricular depolarization), QRS interval (represented ventricular depolarization), QT interval (time corresponding to the beginning of depolarization to repolarization of the ventricles) corrected using Fridericia's formula (QTcF = QT divided by cube root of RR interval) and heart rate (time interval between consecutive heart beats [RR interval]).
Time Frame: Baseline up to Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
percentage of participants | 0

21. Secondary Outcome: Percentage of Participants With Clinically-Significant Radiological Abnormalities
Description: Radiological examination was performed to evaluate presence or signs of infections or pneumonitis.
Time Frame: Baseline up to Month 12
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 52
percentage of participants | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sirolimus
Serious Adverse Events (participants affected / at risk) | 21/52
Other Adverse Events (participants affected / at risk) | 42/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=52)
Escherichia urinary tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia escherichia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Zygomycosis (Infections and infestations) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Generalised oedema (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Spinal pain (General disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 1
Neurological decompensation (Nervous system disorders) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Renal lymphocele (Injury, poisoning and procedural complications) | 1
Transplant rejection (Immune system disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Leg amputation (Surgical and medical procedures) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Blood creatine increased (Investigations) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=52)
Escherichia urinary tract infection (Infections and infestations) | 6
Candidiasis (Infections and infestations) | 5
Onychomycosis (Infections and infestations) | 3
Tinea versicolour (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Acute sinusitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis rotavirus (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 1
Peritonsillitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 5
Lymphocele (Vascular disorders) | 4
Deep vein thrombosis (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Varicose ulceration (Vascular disorders) | 1
Oedema peripheral (General disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 5
Aphthous stomatitis (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 8
Anaemia (Blood and lymphatic system disorders) | 5
Proteinuria (Renal and urinary disorders) | 8
Haematuria (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Weight increased (Investigations) | 3
Blood creatine increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Aphasia (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Trigeminal neuralgia (Nervous system disorders) | 1
Visual field defect NOS (Nervous system disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Visual acuity reduced (Eye disorders) | 2
Conjunctival irritation (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vulvovaginal human papilloma virus infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Mouth injury (Injury, poisoning and procedural complications) | 1
Breast calcifications (Reproductive system and breast disorders) | 1
Haematospermia (Reproductive system and breast disorders) | 1
Panic attack (Psychiatric disorders) | 1
Transplant rejection (Immune system disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Epidermal naevus (Congenital, familial and genetic disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.